CLINICAL TRIAL: NCT06660836
Title: Effect of Digitally Produced Custom Mouthguards on the Awareness and Sports Performance of Child and Adolescent Basketball Players
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Hüseyin Karayılmaz, Professor, Akdeniz University
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: TDH-2024-6739
Record Dates: First submitted 2024-10-22; First posted 2024-10-28 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-10

CONDITIONS: Sports Performance in Children
Keywords: mouthguard; digital workflow; sports performance; protective equipment
MeSH Terms: interventions — Mouth Protectors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Yo-Yo performance test (Other): Participants will undergo the Yo-Yo performance test both while using and not using mouthguards prepared with a digital workflow.
  Interventions: Device: Mouthguard; Other: Performance test

INTERVENTIONS:
Device: Mouthguard — After the participants' records are taken with intraoral scanners, custom mouthguards will be prepared from soft EVA sheets in a dental laboratory setting.
Other: Performance test — Participants will undergo the Yo-Yo performance test both while using and not using mouthguards prepared with a digital workflow.

SUMMARY:
The aim of the study is to investigate the effects of custom mouthguards, prepared using digital workflow, on the sports performance of children and adolescents who play basketball, and to evaluate their views on the use of mouthguards.

Do digitally produced custom mouthguards have an effect on the sports performance of child and adolescent basketball players?

Will the awareness and opinions of child and adolescent basketball players regarding mouthguards be affected?

Participants will:

Undergo the Yo-Yo performance test both while using and not using mouthguards prepared with a digital workflow.

ELIGIBILITY:
Inclusion Criteria:

* Involved in basketball for at least one year,
* Amateur or semi-professional athletes,
* Possession of a health report confirming eligibility for high-activity sports,
* No severe skeletal or dental anomalies,
* Class I occlusion relationship,
* No or mild dental crowding issues,
* No severe nasal deviation that would interfere with sports,
* No prior use of any type of mouthguard,
* Training 4-5 days a week and actively competing in a basketball league.

Exclusion Criteria:

* Individuals with mouth breathing,
* Individuals with a history of adenoid vegetation or enlarged adenoids.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Effects of custom mouthguards on sports performance of child and adolescent basketball players | From enrollment to the end of performance tests, up to 20 weeks
  Effects of custom mouthguards on sports performance of child and adolescent basketball players will be evaluated by a performance test.

SECONDARY OUTCOMES:
Knowledge, awareness, and views on mouthguards | Within 10 minutes after the performance test
  Participants will complete a ...-item questionnaire regarding their knowledge, awareness, and views on mouthguards.

IPD SHARING:
Plan to Share IPD: Undecided